CLINICAL TRIAL: NCT06740058
Title: Bladder Wall Thickness in Symptomatic Urinary Stress Incontinence and Its Correlation with Urodynamics Results. a Retrospective and Prospective Observational Study
Brief Title: Bladder Wall Thickness in Symptomatic Urinary Stress Incontinence and Its Correlation with Urodynamics Results
Acronym: BWT-IUS
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, Professor, IRCCS San Raffaele
Other Study IDs: BWT-IUS
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence , Stress; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This clinical study aims to assess the utility of ultrasonographic bladder wall thickness (BWT) measurement in patients suffering from symptomatic stress urinary incontinence (SUI). SUI is a condition characterized by involuntary leakage of urine during activities that increase intra-abdominal pressure and represents a very frequent disorder impacting women's quality of life. To diagnose SUI more accurately and especially before surgical treatment, patients undergo invasive urodynamic examination. This examination allows us to objectify the presence of any bladder dysfunction and, in particular, to evaluate the presence of detrusor overactivity. Detrusor overactivity is defined as any occurrence of detrusor contraction(s) during filing cystometry. These contractions, which may be spontaneous or provoked, produce a waveform on the cystogram, of variable duration and amplitude and may cause or not urgency symptoms. In absence of any urodynamic detrusor overactivity, the patient may be diagnosed with pure SUI. This is essential to assess before surgical treatment to avoid worsening of symptoms and to decide whether to treat the patient with concomitant pharmacological treatment. On the contrary, ultrasonography offers a non-invasive and accessible approach to evaluate bladder function. This study will involve a cohort of patients with SUI, who will undergo ultrasonographic assessment of BWT and preoperative urodynamic assessment. The objective is to determine whether BWT correlates with the urodynamics results and whether it can predict the presence or absence of detrusor overactivity and confirm the pure stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Women aged > 18 y.o.
3. Women symptomatic for pure or predominant stress incontinence attending the urogynecology outpatient clinic at our institution.
4. Patients undergoing urogynecological standard evaluation for their symptoms, including outpatient gynecological visit and a transvaginal ultrasound.
5. Patients undergoing invasive urodynamic examination for objective assessment of their symptoms or in preparation for possible anti-incontinence surgery.

Exclusion Criteria:

1. Patients with pure or predominant OAB symptomatology
2. Current use of antimuscarinic agents or beta3-agonists (for example Mirabegron)
3. Presence of urological or gynecological cancer.
4. Patients with previous anti-incontinence surgery.
5. Patients with pelvic organ prolapse > II stage.
6. Patients with chronic bladder retention.
7. Patients with neurological diseases that may affect bladder function and urodynamic results.
8. Participants unwilling or unable to give informed consent for participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with pure or prevalent stress urinary incontinence who undergo invasive urodynamic examination
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bladder wall thickness in millimeters (mm) in two different bladder points (dome and trigone) in patients with or without detrusor overactivity at urodynamic assessment | From enrollment to the urodynamic examination that will be performed with 6 months from baseline visit